CLINICAL TRIAL: NCT00783120
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Negative Symptoms in Schizophrenia - a Multicenter Study
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Negative Symptoms in Schizophrenia
Acronym: RESIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Collaborators: University of Göttingen (Other)
Responsible Party: Prof. MD. Peter Falkai, Dept. of Psychiatry and Psychotherapy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RESIS
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Schizophrenia
Keywords: schizophrenia, negative symptoms, TMS, magnetic stimulation
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 10 Hz rTMS of left dorsolateral prefrontal cortex (DLPFC) (15 sessions/3 weeks, 1000 stimuli per session, stimulation intensity 110 % related to the individual resting motor threshold).
  Interventions: Other: Repetitive transcranial magnetic stimulation
- 2 (Sham Comparator): placebo (sham)-rTMS of left DLPFC (15 sessions/3 weeks, 1000 stimuli per session)
  Interventions: Other: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Other: Repetitive transcranial magnetic stimulation — 10 Hz rTMS of left dorsolateral prefrontal cortex (DLPFC) (15 sessions/3 weeks, 1000 stimuli per session, stimulation intensity 110 % related to the individual resting motor threshold); in total 15.000 stimuli.
  Arms: 1
Other: Sham repetitive transcranial magnetic stimulation — placebo (sham)-rTMS of left DLPFC (15 sessions/3 weeks, 1000 stimuli per session; in total 15.000 stimuli
  Arms: 2

SUMMARY:
Schizophrenia is a major psychotic disorder that presents an enormous burden to the patients and their relatives. Despite treatment with second generation antipsychotics, negative symptoms and cognitive impairment often persist and determine an unfavourable course including reduction in life quality. Prefrontal repetitive transcranial magnetic stimulation (rTMS), a promising noninvasive biological technique, applied adjuvant to ongoing antipsychotic treatment was demonstrated to be safe and was associated with improvement in negative symptoms in the majority of the small placebo-controlled trials.

The primary objective of the trial is to investigate the efficacy of high-frequency rTMS (add-on to antipsychotic therapy) in the treatment of negative symptoms in schizophrenia compared to sham stimulation (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Male or female in-patients and out-patients, 18 - 60 years of age
* Diagnostic criteria for schizophrenia according to ICD-10/DSM IV
* PANSS negative sum score > 20 points, 1 of items N1 - N7 (range 1 to 7) ≥ 4 (at least moderate)
* Improvement in PANSS negative sum score less than 10 % in the last 2 weeks prior to study entry, stable antipsychotic medication
* Informed Consent

Exclusion Criteria:

* Clinically relevant psychiatric comorbidity, verbal IQ < 85
* History of epileptic seizures, organic brain disease
* Instable medical comorbidity or condition
* Previous treatment by rTMS
* Factors not compatible with the use of TMS, e.g. cardiac pace makers or other metallic implants, pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Improvement in negative symptoms (baseline vs. day 21, PANNS negative sum score) | 105 Days

SECONDARY OUTCOMES:
efficacy on cognition, EPS, neuroplasticity (sMRI/MRS), depression, life quality and social function | 105 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Falkai, Prof MD., Study Director — Dept. of Psychiatry and Psychotherapy, University Hospital of the Georg-August-University Göttingen
Locations (3):
- Germany (3):
  - Department of Psychiatry and Psychotherapy, University of Regensburg, Regensburg, Bavaria
  - Dept. of Psychiatry and Psychotherapy, University Hospital of the Georg-August-University Göttingen, Göttingen, Lower Saxony
  - Department of Psychiatry, Heinrich-Heine University Hospital, Düsseldorf, North Rhine-Westphalia

REFERENCES:
- [Derived] Koutsouleris N, Wobrock T, Guse B, Langguth B, Landgrebe M, Eichhammer P, Frank E, Cordes J, Wolwer W, Musso F, Winterer G, Gaebel W, Hajak G, Ohmann C, Verde PE, Rietschel M, Ahmed R, Honer WG, Dwyer D, Ghaseminejad F, Dechent P, Malchow B, Kreuzer PM, Poeppl TB, Schneider-Axmann T, Falkai P, Hasan A. Predicting Response to Repetitive Transcranial Magnetic Stimulation in Patients With Schizophrenia Using Structural Magnetic Resonance Imaging: A Multisite Machine Learning Analysis. Schizophr Bull. 2018 Aug 20;44(5):1021-1034. doi: 10.1093/schbul/sbx114. PMID 28981875
- [Derived] Hasan A, Wobrock T, Guse B, Langguth B, Landgrebe M, Eichhammer P, Frank E, Cordes J, Wolwer W, Musso F, Winterer G, Gaebel W, Hajak G, Ohmann C, Verde PE, Rietschel M, Ahmed R, Honer WG, Dechent P, Malchow B, Castro MFU, Dwyer D, Cabral C, Kreuzer PM, Poeppl TB, Schneider-Axmann T, Falkai P, Koutsouleris N. Structural brain changes are associated with response of negative symptoms to prefrontal repetitive transcranial magnetic stimulation in patients with schizophrenia. Mol Psychiatry. 2017 Jun;22(6):857-864. doi: 10.1038/mp.2016.161. Epub 2016 Oct 11. PMID 27725655
- [Derived] Wobrock T, Guse B, Cordes J, Wolwer W, Winterer G, Gaebel W, Langguth B, Landgrebe M, Eichhammer P, Frank E, Hajak G, Ohmann C, Verde PE, Rietschel M, Ahmed R, Honer WG, Malchow B, Schneider-Axmann T, Falkai P, Hasan A. Left prefrontal high-frequency repetitive transcranial magnetic stimulation for the treatment of schizophrenia with predominant negative symptoms: a sham-controlled, randomized multicenter trial. Biol Psychiatry. 2015 Jun 1;77(11):979-88. doi: 10.1016/j.biopsych.2014.10.009. Epub 2014 Oct 23. PMID 25582269
- [Derived] Cordes J, Falkai P, Guse B, Hasan A, Schneider-Axmann T, Arends M, Winterer G, Wolwer W, Ben Sliman E, Ramacher M, Schmidt-Kraepelin C, Ohmann C, Langguth B, Landgrebe M, Eichhammer P, Frank E, Burger J, Hajak G, Rietschel M, Wobrock T. Repetitive transcranial magnetic stimulation for the treatment of negative symptoms in residual schizophrenia: rationale and design of a sham-controlled, randomized multicenter study. Eur Arch Psychiatry Clin Neurosci. 2009 Nov;259 Suppl 2:S189-97. doi: 10.1007/s00406-009-0060-y. PMID 19876678